CLINICAL TRIAL: NCT03003689
Title: Randomized Clinical Trial Assessing the Clinical Outcomes and Recolonization Patterns Following Scaling and Root Planing With and Without Using Er.YAG Laser in Chronic Periodontitis Patients
Brief Title: Effects of Scaling and Root Planing With and Without Er:YAG Laser in Chronic Periodontitis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tufts University School of Dental Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12321
Record Dates: First submitted 2016-12-09; First posted 2016-12-28 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Chronic Periodontitis
Keywords: Scaling and Root Planing; Er:YAG
MeSH Terms: conditions — Chronic Periodontitis | interventions — Tooth Exfoliation; Root Planing; Lasers, Solid-State

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Scaling and Root Planing (Active Comparator): Hand instruments + ultrasonic scaler
  PD, CAL, plaque index and gingival bleeding index will be measured at baseline, 6 weeks and 3 months. Microbial load will be measured at baseline and 3 months.
  Interventions: Procedure: Scaling and Root Planing
- Scaling and Root Planing + Er:YAG Laser (Experimental): Er:YAG Laser, hand instruments + ultrasonic scaler
  PD, CAL, plaque index and gingival bleeding index will be measured at baseline, 6 weeks and 3 months. Microbial load will be measured at baseline and 3 months.
  Interventions: Procedure: Scaling and Root Planing; Device: Er:YAG Laser

INTERVENTIONS:
Procedure: Scaling and Root Planing — Standard of care scaling and root planing using hand instruments and ultrasonic scaler
Device: Er:YAG Laser — Er:YAG laser as an adjunct therapy to standard of care scaling and root planing using hand instruments and ultrasonic
  Arms: Scaling and Root Planing + Er:YAG Laser

SUMMARY:
Dental bacterial plaque is the most frequent modifiable finding in patients with periodontal (gum) diseases. Many studies have provided evidence that mechanical removal of dental plaque is critical for improving the periodontal health. The standard initial treatment of periodontitis (gum disease) is to remove plaque and calculus form the teeth and root structures using sclaing and root planing (SRP). Typically hand instruments and an ultrasonic scaler are used for SRP

While this method removes some of the bacteria that leads to periodontitis, microorganisms are not completely eliminated through SRP. Studies have shown that after 3 months, the bacteria initially present prior to scaling and root planing had recolonized. In order to prevent recurrence of periodontitis, it is recommended that oral bacteria be kept at low levels.

When used at the proper wave length, dental lasers have been shown to effectively removes calculus, without damaging surrounding tissue. The Er:YAG laser has been FDA-approved for the use of scaling and root planing in Dentistry. While studies on the Er:YAG laser have shown that it is effective in removing calculus and preserving the tooth root structure, there is no consensus of the level of calculus removal. The Er:YAG laser may also be more effective in removing microbial bacteria than SRP with hand instruments and ultrasonic scaler.

The purpose of this study is to evaluate the effectiveness of the Er:YAG laser, as an adjunct to scaling and root planing, in removing microbial bacteria. Participants with chronic periodontitis will be randomized to have one quadrant undergo scaling and root planing using hand instruments and ultrasonic scaler alone, while a second quadrant will receive the same treatment, with the addition of the Er:YAG laser. Outcomes studies will be traditional periodontal clinical parameters at 6 weeks and 3 months after treatment. Microbial cultures will be performed at baseline and 3 months to compare survival and re-population by periodontal microorganisms.

DETAILED DESCRIPTION:
Primary Aim: The primary aim of this study is to evaluate the efficacy of Er:YAG laser as an adjunct to mechanical scaling and root planing periodontal therapy by comparing probing depth and clinical attachment levels.

Secondary aim: The secondary aim of this study is to evaluate the efficacy of Er:YAG laser as an adjunct to mechanical scaling and root planing periodontal therapy by comparing gingival bleeding index and plaque index.

Tertiary aim: The tertiary aim of this study is to compare the microbial outcomes of mechanical periodontal therapy alone vs. mechanical therapy combined followed with Er:YAG laser therapy at the same time.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in the Post-Graduate Periodontology Clinic at Tufts University School of Dental Medicine (TUSDM)
* Recent (within the past 30 days) diagnosis of moderate to severe chronic periodontitis in at least two quadrants according to the Armitage Classification
* Have had full mouth and vertical bite-wing series of diagnostic radiographs exposed at TUSDM within 6 months preceding entry of the study as a standard of care
* Have a treatment plan made by the original provider and certified by the PI based on the working diagnosis, presenting etiology, and the predicted therapeutic outcomes of the case (prognosis).
* Each of the two selected quadrants should have at least 5 teeth including the canine, first premolar and second premolar in contact with at least one tooth that has ≥ 5 mms and ≤ 9 mms probing depths with bleeding on probing.

Exclusion Criteria:

* Participants must not have had mechanical debridement or any other professional periodontal therapy within 6 months preceding entering the study
* Participants with significant chronic oral soft tissue pathology (lichen planus, Benign Mucous Membrane Pemphigoid, Steven Johnson's Syndrome, Sjogren's Syndrome, etc.) which might affect host response to the presence of bacteria.
* Participants with fixed appliances or partial dentures, to standardize the effect of the treatment since they are plaque retentive.
* Participants who smoke tobacco
* Participants who require prophylactic antibiotics prior to dental treatment
* Participants who have taken systemic antibiotic medications within the previous 6 months
* Participants with uncontrolled systemic conditions or disease such as diabetes and immunological disorders
* Participants with known drug allergies or known adverse effects following the use of oral hygiene products.
* Participants who are pregnant or lactating
* Teeth with grade III mobility or teeth with hopeless prognosis indicated for extraction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2017-04-20 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Change in Probing Depth | Up to 3 months
  Differences in pocket depth reduction between laser treatment and control groups will be analyzed with a linear mixed effects model. Four sites (mesiolingual, mesiobuccal, distolingual, and distobuccal) per tooth will be averaged and used in the linear mixed effects model. Normality of the data will be assessed graphically and with the Shapiro-Wilk test.
Change in Clinical Attachment Levels | Up to 3 months
  Differences in attachment gain between laser treatment and control groups will be analyzed with a linear mixed effects model. Four sites (mesiolingual, mesiobuccal, distolingual, and distobuccal) per tooth will be averaged and used in the linear mixed effects model. Normality of the data will be assessed graphically and with the Shapiro-Wilk test.

SECONDARY OUTCOMES:
Change in Gingival Bleeding Index | Up to 3 months
  The gingival bleeding index (the number of bleeding sites divided by the total number of sites) will be calculated. Statistical significance between the two groups' gingival bleeding index will be determined with generalized estimating equations.
Change in Plaque Index | Up to 3 months
  The plaque index (the number of surfaces with plaque divided by the total number of surfaces) will be calculated. Statistical significance between the two groups' plaque index will be determined with generalized estimating equations.
Change in microbial load, measured in Colony Forming Units (CFUs) | baseline, 3 months
  Microbial load will be measured by the total number of cultivable bacteria measured by total viable colony forming units (CFUs) on non-selective and selective media. Percent cultivability of periodontal pathogens will be measured by number of pathogen specific CFUs in proportion to total cultivability.
  Differences in microbial load will be investigated with the paired t-test. If the assumption of normality is unmet, the Wilcoxon rank-sum test will be used instead.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Hawley, DDS, MS, PhD, Principal Investigator — TUSDM
Locations (1):
- Tufts University School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No